CLINICAL TRIAL: NCT07351136
Title: Novel Diagnostic and Prognostic Predictors in Fabry Cardiomyopathy: Proof of Concept in a Rare Disease
Acronym: FABRyCar
Status: Not yet recruiting | Type: Observational
Sponsor: Núcleo de Apoio à Investigação Clínica - FMUP (Other)
Collaborators: Universidade do Porto (Other); SOFIE (Industry); GE Healthcare (Industry)
Responsible Party: Sponsor-Investigator, Núcleo de Apoio à Investigação Clínica - FMUP, Elisabete Martins, Universidade do Porto
Organization: Universidade do Porto (Other)
Other Study IDs: FABRyCar
Record Dates: First submitted 2026-01-09; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-10

CONDITIONS: Fabry Disease
Keywords: Fabry Disease; FAPI
MeSH Terms: conditions — Fabry Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- adults with Fabry disease
  Interventions: Procedure: PET scan of 68Ga-FAPI

INTERVENTIONS:
Procedure: PET scan of 68Ga-FAPI — To assess myocardial fibroblast activation, all enrolled patients will undergo positron emission tomography/computed tomography (PET/CT) imaging using the radiotracer [68Ga]Ga-FAPI. This tracer binds selectively to the fibroblast activation protein (FAP), expressed predominantly in activated cardiac fibroblasts involved in pathological myocardial remodelling.

SUMMARY:
In this work, we address the understanding of the signaling pathways involved in cardiac remodeling in human SCD through molecular imaging analysis with a fibrosis marker. Furthermore, we emphasize characterizing the cardiac remodeling process by analyzing proteomic data from SCD myocardial biopsies and by analyzing the profile of microRNAs associated with hypertrophic cardiomyopathy and their diagnostic and prognostic value.

DETAILED DESCRIPTION:
The objective of this work is to explore the cardiac PET/CT imaging characteristics of cardiac fibroblast activation protein inhibitor (FAPI) and its relationship with the risk of sudden cardiac death (SCD) associated with myocardial fibrosis in SCD.

We also aim to deepen our understanding of the signaling pathways involved in SCD cardiac remodeling by comparing imaging data with proteomic and microRNA data.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, over 18 years of age;
* Diagnosis of Fabry disease

Exclusion Criteria:

* Refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients, over 18 years of age with diagnosis of Fabry disease
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Identify and validate novel molecular biomarkers and pathophysiological mechanisms of FD cardiomyopathy, focusing on myocardial fibrosis, inflammation, and cardiac remodelling | All enrolled patients will undergo PET/CT imaging using the radiotracer [68Ga]Ga-FAPI. This procedure will be done from October 2025 to January 2026. The data analysis will be done from January 2026 to April 2026
  The primary objective includes:
  * Proteomic and metabolomic profiling of myocardial biopsies from FD patients versus controls.
  * Circulating microRNA (miRNA) analysis in plasma samples from HCM and FD patients to define diagnostic/prognostic miRNA signatures.
  * Evaluation of fibroblast activation using [68Ga]Ga-FAPI PET/CT imaging and its association with myocardial fibrosis and sudden cardiac death risk scores.
  * Correlation of molecular findings with cardiac imaging and standard biomarkers (NT-proBNP, troponin).